CLINICAL TRIAL: NCT03404947
Title: Substrate Metabolism During 2 Hours of Moderate Intensity Exercise Following Ingestion of Ethanol in Man
Brief Title: Substrate Metabolism During Exercise Following Ingestion of Ethanol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Betts, Principal Investigator, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ETOH-hs565
Record Dates: First submitted 2017-12-05; First posted 2018-01-19 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Exercise Metabolism Following Ethanol Ingestion
Keywords: Exercise; Metabolism; Nutrition
MeSH Terms: conditions — Motor Activity | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethanol (Experimental): Participants will ingest ethanol (in the form of 40% ethanol) at an ingestion rate of 0.1 grams/kg lean body mass/hour in a solution with water.
  Interventions: Dietary Supplement: Ethanol
- No Ethanol (No Intervention): Participants will ingest a volume matched beverage of water only.

INTERVENTIONS:
Dietary Supplement: Ethanol — For one exercise session, participants will be asked to ingest a quantity of ethanol (in the form of vodka) sufficient to maximally stimulate liver alcohol metabolism.
  Arms: Ethanol

SUMMARY:
This study will investigate how ethanol (pure alcohol) influences carbohydrate and fat metabolism during prolonged, moderate intensity exercise. Participants will perform two bouts of cycling exercise with or without prior ingestion of ethanol, in a randomised order, separated by one week.

DETAILED DESCRIPTION:
Very little research has investigated the influence of ethanol on metabolism during prolonged exercise. Evidence suggests that delivery of fat to the working muscles during exercise may be limited with ethanol and therefore this may shift the relative proportions of energy derived from muscle stores of carbohydrate as a result (Jorfeldt & Juhlin-Dannfelt, 1976).

The current study aims to investigate how a small-moderate dose of ethanol influences where energy is derived from during a prolonged bout of moderate intensity cycling exercise.

Participants will visit the lab on three occasions, once for preliminary measurements of fitness and body composition, and twice for the experimental bouts of exercise. Body composition will be assessed using a dual-energy x-ray absorptiometry (DEXA) scan, which will measure lean mass, fat mass, and bone mineral density. Participants will then perform an incremental maximal oxygen uptake test to determine intensity for the experimental bouts of exercise.

The two experimental bouts of exercise include cycling on an exercise bike for 2 hours at 55% of their maximal oxygen uptake (i.e. fitness) following 1 hours rest. This will be performed under two conditions: with and without ethanol ingestion. Pre and post exercise muscle biopsies will be collected to assess muscle metabolism, with regular blood samples and expired breath samples being collected to further investigate fuel delivery and use by the working tissues. The experimental bouts of exercise will be performed 1 week apart in a randomised order.

ELIGIBILITY:
Inclusion Criteria:

* Habitual alcohol consumer (average 1-14 units per week)
* BMI 18.5 - 29.9 kg/m2
* Be able to attend the laboratory and willing to participate in necessary protocols
* Be willing to undertake the durations of the exercise protocol (2 hours) ]
* Have the capacity and willingness to provide informed consent (oral and written)

Exclusion Criteria:

* Non-or excessive alcohol drinkers (0 or >14 units per week)
* History of substance abuse
* Habitual/previously habitual smokers
* BMI >30.0 kg/m2
* Experience contraindications to the administration of the proposed anaesthetic (Lidocaine Hydrochloride)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Change in muscle glycogen content | Change in muscle glycogen content over 2 hours of moderate intensity cycling exercise
  Muscle biopsy and subsequent biochemical analysis
Blood glucose concentration | Blood samples will be taken every 15 minutes during rest and the first hour of exercise, they will be taken every 30 minutes in the second hour of exercise.
  Venous blood samples will be taken and biochemically analysed for blood glucose concentration.
Blood non-esterified fatty acid (NEFA) concentration | Blood samples will be taken every 15 minutes during rest and the first hour of exercise, they will be taken every 30 minutes in the second hour of exercise.
  Venous blood samples will be taken and biochemically analysed for NEFA concentration.

SECONDARY OUTCOMES:
Blood ethanol concentration | Blood samples will be taken every 15 minutes during rest and the first hour of exercise, they will be taken every 30 minutes in the second hour of exercise.
  Venous blood samples will be taken and biochemically analysed for blood ethanol concentration.
Blood lactate concentration | Blood samples will be taken every 15 minutes during rest and the first hour of exercise, they will be taken every 30 minutes in the second hour of exercise.
  Venous blood samples will be taken and biochemically analysed for blood lactate concentration.
Carbohydrate Oxidation | Expired breath samples will be collected at baseline before beverage consumption and again after 1 hours rest. Samples will collected every 15 minutes during the first hour of exercise and every 30 minutes during the second hour
  Carbohydrate oxidation will be determined through indirect calorimetry via the douglas bag technique.
Fat Oxidation | Expired breath samples will be collected at baseline before beverage consumption and again after 1 hours rest. Samples will collected every 15 minutes during the first hour of exercise and every 30 minutes during the second hour
  Fat oxidation will be determined through indirect calorimetry via the douglas bag technique.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Smith, Principal Investigator — University of Bath; James Betts, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jorfeldt L, Juhlin-Dannfelt A. The influence of ethanol on human splanchnic and skeletal muscle metabolism during exercise. Scand J Clin Lab Invest. 1977 Nov;37(7):609-18. doi: 10.3109/00365517709100653. No abstract available. PMID 594641
- [Background] Juhlin-Dannfelt A, Ahlborg G, Hagenfeldt L, Jorfeldt L, Felig P. Influence of ethanol on splanchnic and skeletal muscle substrate turnover during prolonged exercise in man. Am J Physiol. 1977 Sep;233(3):E195-202. doi: 10.1152/ajpendo.1977.233.3.E195. No abstract available. PMID 910908
- [Background] Juhlin-Dannfelt A, Jorfeldt L, Hagenfeldt L, Hulten B. Influence of ethanol on non-esterified fatty acid and carbohydrate metabolism during exercise in man. Clin Sci Mol Med. 1977 Sep;53(3):205-14. doi: 10.1042/cs0530205. No abstract available. PMID 913043